CLINICAL TRIAL: NCT02628756
Title: Endometrial Injury Does Not Improve Pregnancy Rates in Women With Unexplained Infertility
Brief Title: Endometrial Injury in Women With Unexplained Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura Integrated Fertility Center (Other)
Responsible Party: Principal Investigator, Tarek Shokeir, Prof. Obstetrics & Gynecology, Mansoura Integrated Fertility Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS/490
Record Dates: First submitted 2015-12-08; First posted 2015-12-11 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Unexplained Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endometrial injury (Experimental): Hysteroscopic-guided endometrial injury (Karl Storz, Tuttlingen, Germany).
  Interventions: Procedure: Endometrial injury

INTERVENTIONS:
Procedure: Endometrial injury — Office hysteroscopy (Karl Storz, Tuttlingen, Germany)

SUMMARY:
Women between 18-39 years old who had been infertile (primary or secondary) for at least 1 year were recruited. In a parallel assignment eligible participants were randomized to receive either a single, site-specific endometrial injury guided by hysteroscopy (Study group) or no intervention (Control group). Natural cycle folliculometry + timed sexual intercourse were offered for all participants for the ongoing and the immediate 2 concecutive cycles. Clinical pregnancy rates were the primary outcome and miscarriage rates were the secondary outcome measures.

DETAILED DESCRIPTION:
A single site-specific hysteroscopic injury procedure (Snip) will be performed using an office hysteroscopy (Karl Storz, Germany). By means of vaginoscopy, a 2.9 mm. continuous-flow diagnostic hysteroscope with a 5 Fr. working-channel is guided through the cervical canal with normal saline as distension medium, with flow manually regulated through the key of the hysteroscopic sheath.

The examination of the uterine cavity begins by observing its regularity, paying special attention to the presence of intrauterine malformations or morphologic alterations such as submucous myomas, or uterine septa. Subsequently, A claw forceps will be introduced through a 2.2 mm working channel, and will be used to generate a local injury on the upper posterior endometrium (Endometrial Snip) at midline 10-15 mm from the fundus on D4 to D7 of the ongoing menstrual cycle. The depth and width of the injured site will be about 2x2 mm (i.e a single bite of the claw forceps). No premedications, antibiotics or hemostatics will be given after the procedure.

Natural cycle folliculometry + timed sexual intercourse will be offered for all participants for the ongoing and the immediate subsequent cycles. Once the leading ovarian follicle will reach a size of at least 16 mm, 10,000 IU of hCG will be administered to trigger ovulation.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 39 years old.
2. Normal HSG and/or diagnostic laparoscopy.
3. Normal seminal profile.
4. Regular ovulation confirmed by mid-luteal progesterone.
5. Normal TVS criteria.

Exclusion Criteria:

1. Uterine fibroid.
2. Pelvic endometriosis.
3. Irregular menstruation.
4. Ovarian cysts.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rates (PR) | Three consecutive months

SECONDARY OUTCOMES:
Miscarriage rates | Three consecutive months

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Shokeir, M.D., Principal Investigator — Mansoura University Hospital, Mansoura Faculty of Medicine